CLINICAL TRIAL: NCT02210403
Title: The Influence of tDCS on the Arm and Hand Function in Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: S54797
Record Dates: First submitted 2014-07-24; First posted 2014-08-06 (Estimated); Last update posted 2023-03-28 (Actual); Status verified 2013-02

CONDITIONS: Transcranial Direct Current Stimulation; Cerebrovascular Accident (CVA)
MeSH Terms: conditions — Stroke | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Upper limb motor function training + tDCS (Active Comparator): Bi-hemispheric tDCS with motor function training
  Interventions: Device: transcranial direct current stimulation (tDCS)
- upper limb motor function training + sham tDCS (Sham Comparator): sham tDCS with motor function training
  Interventions: Device: transcranial direct current stimulation (tDCS)

INTERVENTIONS:
Device: transcranial direct current stimulation (tDCS)

SUMMARY:
The purpose of this study is to determine whether tDCS in combination with motor training can improve hand and arm function in stroke patients.

ELIGIBILITY:
Inclusion Criteria:

* Stroke patients onset > 6 months
* First ever stroke
* Decreased hand and arm function
* Mini Mental State Examination (>24)

Exclusion Criteria:

* Depression
* Pregnancy
* Alcohol abuse
* Aneurysm clips
* Pacemaker
* Neurostimulator
* Implemented defibrillator
* Magnetically activated implant or device
* implemented pump
* Spinal cord simulator
* Implemented hearing aid
* Artificial or prosthetic limb
* Metal parts in the body
* Any external or internal metal
* Artificial heart valve
* Other implants
* History of brain surgery
* Migraine
* Family history of Epilepsy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2013-04-18; Primary Completion 2014-09-28 (Actual); Study Completion 2014-09-28 (Actual)

PRIMARY OUTCOMES:
Change of Fugl-Meyer assessment (FMA) score | Change from baseline in FMA score on the 3rd intervention day; change from baseline in FMA score at 1 week post intervention

SECONDARY OUTCOMES:
Change of Modified Ashworth scale (MAS) | Change from baseline in MAS scale on the 3rd intervention day; change from baseline in MAS scale at 1 week post intervention

OTHER OUTCOMES:
Change of motor task performance | Change from baseline motor task performance on the 3rd intervention day, and change from baseline in motor task performance at 1 week post intervention

CONTACTS AND LOCATIONS:
Locations (1):
- K U Leuven, Leuven, Belgium

REFERENCES:
- [Derived] Zhang X, Meesen R, Swinnen SP, Feys H, Woolley DG, Cheng HJ, Wenderoth N. Combining muscle-computer interface guided training with bihemispheric tDCS improves upper limb function in patients with chronic stroke. J Neurophysiol. 2024 Jun 1;131(6):1286-1298. doi: 10.1152/jn.00316.2023. Epub 2024 May 8. PMID 38716555
- [Derived] Elsner B, Kugler J, Pohl M, Mehrholz J. Transcranial direct current stimulation (tDCS) for improving activities of daily living, and physical and cognitive functioning, in people after stroke. Cochrane Database Syst Rev. 2020 Nov 11;11(11):CD009645. doi: 10.1002/14651858.CD009645.pub4. PMID 33175411